CLINICAL TRIAL: NCT05972031
Title: EMBOSS: Reach and Effect of a Person-centred Integrated-care Approach for Chronic Diseases and MultimorBidity in Patients of Low sOcio- Economic StatuS in General Practice
Brief Title: EMBOSS A Person-centred Integrated-care for Chronic Diseases in Patients of Low Socio Economic Status
Acronym: EMBOSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-15786
Record Dates: First submitted 2023-02-06; First posted 2023-08-02 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-02

CONDITIONS: Chronic Condition; Chronic Conditions, Multiple
Keywords: Primary care; Person-centered; Integrated-care; Health literacy; Health disparities; Socio-economic status; General practice
MeSH Terms: conditions — Chronic Disease; Multiple Chronic Conditions

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Person-centred integrated care intervention (Experimental): The core of the person-centered approach is a cyclical process and for EMBOSS developed for patients with low SES. The practice nurse in the GP will act as case manager and can consult other health providers. The first step in the intervention is assessing the integral health status of the patient (health across multiple domains), using a visual conversation tool. The second step is discussing the results with the patient. Personal goals are formulated in the third step. In the fourth step, the healthcare professional and patient will choose through shared-decision making the most appropriate interventions and support to achieve these goals, which are documented in a personal plan. Next, referrals are made if necessary and the treatment is started. An evaluation is planned and carried out. All practices in the EMBOSS intervention group will be trained by Pharos on how to recognize and provide GDM to low SES patients using appropriate communication skills and the specific tools.
  Interventions: Behavioral: Person-centred integrated care intervention
- Usual care (No Intervention): Practices in the control group provide care as usual, which consists of the SDM programmes according to the national care standards and General Practice guidelines (NHG) for DM2, COPD and CVD. According to these protocolised programmes, patients with COPD, CVD or DM2 visit their general practice at a standard frequency per year (1 - 4 times) and standard monitoring measurements and topics are discussed.
  The practices that are randomised to the control group will not receive any additional training related to this study.

INTERVENTIONS:
Behavioral: Person-centred integrated care intervention — See arm description.
  Other Names: Usual care
  Arms: Person-centred integrated care intervention

SUMMARY:
People of low socio economic status (SES) more often than others suffer from chronic diseases like diabetes mellitus, chronic obstructive pulmonary disease (COPD), or coronary diseases. Compared to others People of low SES more often have to deal with multiple diseases (multimorbidity) and experience worse health outcomes. The health literacy of people of low SES is often low. Current chronic disease management programs focus on reducing the burden of a single disease by prescribing medication, protocoled monitoring routines, or lifestyle advice.

However, the effectiveness of these interventions is low in people with low SES, as the interventions insufficiently take into account the specific problems and needs of this (multimorbid) population. A person-centered and integrated-care approach, that puts the patient at the center of care instead of the disease and in which care is tailored to the individual patient with chronic disease(s), seems to be more appropriate, but only when low SES people are closely involved in the development, testing, and evaluation of such an approach. Also, certain preconditions should be met, such as training of specific knowledge and skills of the healthcare professionals involved.

In the EMBOSS project, the investigators will develop, test, evaluate, and implement a person-centered integrated-care approach for and in close collaboration with people with low SES who have one or more chronic diseases. Thus, the EMBOSS study will have the potential to reducing health disparities in this group, to broadening the action perspectives of general practitioners and practice nurses for an increasing diverse patient population and to a better fit of lifestyle interventions in people of low SES.

DETAILED DESCRIPTION:
In the Netherlands, 28% of the population is lowly educated, i.e. the level of education is MBO1 (secondary vocational education) or lower, which is the main indicator of low socioeconomic status. Low-educated people suffer 2-4 times more often than high-educated people from diabetes mellitus, COPD, coronary disease (often in combination) and of the risk factors contributing to these diseases. The healthy life-expectancy for low educated people is 14 years shorter, the health outcomes are worse (more complications of cardiovascular diseases and diabetes), because of high levels of chronic stress due to challenging living circumstances, negatively influencing self-confidence and executive functions, limited health and digital literacy - all determinants of effective self-management. Most people with chronic diseases are being cared for in general practice (GP). However, professionals in GP often struggle with the care for low-educated patients, experiencing difficulties in recognizing patients with low (health) literacy, and in adapting communication and advice to the needs of this group. Low-educated patients more often visit the GP, and are more often referred to costly secondary care.

Many interventions for chronic diseases fail to show effectiveness in low-SES groups. The reasons are multiple:

1. materials and procedures used are too complicated,
2. daily survival sets different priorities,
3. communication and approach by healthcare professionals don't suit the needs and skills of this population, actions or materials are too expensive.

Effectiveness of interventions can be improved by involving low-SES patients in the development and by training healthcare professionals. Low-educated patients should be explicitly recruited in intervention evaluation studies as this population is underrepresented in clinical studies, which impedes generalizability of results. Chronic care for patients with diabetes mellitus type 2 (DM2), COPD and/or cardiovascular diseases (CVD) in GP is carried out through disease management programmes. However, major limitations of these programmes are that it focused on a single disease, while half of the patients suffers from multimorbidity. Also, the programmes do not truly reflect the needs of patients who experience this disease management as fragmented with too little attention for the partienst personal context. Therefore, a more generic disease management (GDM) programme including a person-centred and integrated-care (PC-IC) approach seems to be a promising strategy. Such an approach puts the patient at the centre of care, tailoring chronic care to the individual's needs and addressing all the issues important to him. It starts with a comprehensive biopsychosocial assessment of all relevant problems. Subsequently, a personalised treatment plan is made with individualised goals, actions and professionals involved. The programme responds to the needs and context of the 'whole' patient to provide the right care in the right place at the right time. It supposes to stimulate patient's self-management.

Currently, in the Netherlands, some regional projects with GDM programmes and PC-IC approaches are running, of which 'OPTIMA FORMA' may be the best known. This project started in 2018 and consists of three stages in which a GDM programme including a PC-IC approach is developed, tested and evaluated in three large Dutch primary care cooperatives, i.e Nijmegen, Arnhem, and Doetinchem. However, in 'OPTIMA FORMA' as in other ongoing projects, there is no specific attention for or involvement of people with low SES. This will obviously reduce the effectiveness of this approach in low SES patients, as one third of the population with chronic diseases consists of patients with low SES. The investigators there is an urgent need for PC-IC interventions that specifically address the needs of low SES population in order to be effective. Therefore, the investigators supported the three primary care cooperatives who participate in OPTIMA FORMA with the development of a GDM programme specifically for low SES patients. With help from patients with low SES and the healthcare professionals of the low SES patient, the investigators collected information on experiences, facilitators, and barriers from the previously conducted pilot study of OPTIMA FORMA PHASE2 (CMO 2021-8106).

The investigators used this information in co-creation sessions with patients with low SES and healthcare professionals to adjust the OPTIMA FORMA programme to a GDM programme that better suits the needs of low SES patients (EMBOSS programme).

The hypothesise off the EMBOSS programme will not only result in better outcomes of care in this group (and thus decreasing socio-economic health disparities), but also to a more effective role of GPs and practice nurses with more work satisfaction and less workload. In the current study our primary research question is:

What is the effectiveness of the EMBOSS intervention, i.e. a GDM programme including a PC-IC approach developed with and for low SES people with one or more chronic diseases compared to care as usual, i.e. SDM programmes for DM2, COPD and/or CVD in general practice? The investigators will perform a cluster randomized controlled trial with a follow-up time of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in any of the single disease management programmes (usual care) for DM2, COPD, asthma or CVD

Exclusion Criteria:

* Limited life expectancy (less than 3 months)
* Patients with high level of SES (or educational level > MBO2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2023-01-29 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
patient-reported health-related quality of life Physical Health | 12 months
  Global Physical Health [Time Frame: Baseline, 6 months, 12 months] Physical aspect of health-related quality of life as measured by the PROMIS-Global 10 instrument (T-scores; higher T-score indicates better physical aspect of HrQoL) Promis 10 is a patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales.
patient-reported health-related quality of life Mental health | 12 months
  Global Mental Health [Time Frame: Baseline, 6 months, 12 months] Mental aspect of health-related quality of life as measured by the PROMIS-Global 10 instrument (T-scores; higher T-score indicates better mental aspect of HrQoL) Promis 10 is a patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales.
Patient-experienced quality of care | 12 months
  atient-experienced quality of care [Time Frame: Baseline, 6 months, 12 months] Person-centredness of care as measured by the Person Centred Coordinated Care Experience Questionnaire (P3CEQ) instrument; minimum score 0, maximum score 30, higher score equals better P3CE.

SECONDARY OUTCOMES:
Patient activation as measured by PAM | Baseline, 6 months, 12 months
  Patient activation as measured by the Patient Activation Measure instrument; minimum 0, maximum 100, higher score equals better patient activation.
Health-related quality of life as measured by the EQ-5D-5L instrument | Baseline, 6 months, 12 months
  Health-related quality of life as measured by the EQ-5D-5L instrument; minimum 0, maximum 1, higher score equals better HrQoL
BMI | Baseline, 6 months, 12 months
  Combined length and weight according to general practice data (registered for normal care)
HbA1c | Baseline, 6 months, 12 months
  according to general practice data
Blood glucose | Baseline, 6 months, 12 months
  according to general practice data
Blood LDL-cholesterol | Baseline, 6 months, 12 months
  according to general practice data
Systolic and diastolic blood pressure | Baseline, 6 months, 12 months
  according to general practice data
Positive affect of healthcare providers | Baseline, 6 months, 12 months
  Satisfaction with job according to selection of MAS-GZ instrument (minimum 8, maximum 40, higher score indicates higher positive affect)
Experience of healthcare providers | Baseline, 6 months, 12 months
  Satisfaction with job according to selection of CO-PILOT instrument (minimum 1, maximum 10, higher score is better experience of healthcare providers)

CONTACTS AND LOCATIONS:
Locations (1):
- RadboudUMC, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided